CLINICAL TRIAL: NCT03264430
Title: Adding Ketamine to Low Dose Bupivacaine in Saddle Block for Perianal Surgery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Esam Eldin Mohamed Abdalla (Other)
Responsible Party: Sponsor-Investigator, Esam Eldin Mohamed Abdalla, Clinical Professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17100219
Record Dates: First submitted 2017-05-29; First posted 2017-08-29 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Perianal Fistula; Hemorrhoids
Keywords: Perianal fistula; Hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Ketamine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The ketamine group (Active Comparator): The ketamine group will receive intrathecal bupivacaine (7.5 mg) in 1.5 ml (Marcaine, Astra Zeneca, France, 0.5%) and ketamine (25mg) in 0.5 ml (Ketam, EIPICO, Egypt, 50 mg/mL),. Total volume is 2 ml will injected
  Interventions: Drug: Ketamine; Drug: bupivacaine
- The control group (Placebo Comparator): group will receive only intrathecal bupivacaine (7.5 mg) in 1.5 ml plus 0.5ml normal saline to achieve total volume of 2 ml.
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: Ketamine — an antagonist of the NMDA receptor
  Other Names: ketalar
  Arms: The ketamine group
Drug: bupivacaine — local anaesthetic
  Other Names: marcaine 0.5 %

SUMMARY:
Evaluation of the anesthetic quality and analgesic efficacy of adding ketamine to intrathecal bupivavaine in selective saddle block for perianal surgery.

DETAILED DESCRIPTION:
This study will be carried out in Assiut University Hospitals, General Surgery Operative room and Post Anaesthesia Care Unit (PACU).

This study will include 60 adult participants (ASA I&II) scheduled for minor perianal surgery (perianal fistula, haemorrhoids or both). After approval of ethics committee and written informed consent will be obtained from the participants.

Investigators will exclude participants with classic contraindications to spinal block, pre-existing systemic disease (such as cardiovascular, respiratory or renal diseases), coagulopathy and participants taking any medications that could influence the haemodynamic response.

The selected participants will be divide into two groups (30 participants for each group), ketamine group and placebo (control) group.

The ketamine group will receive intrathecal bupivacaine (7.5 mg) in 1.5 ml (Marcaine, Astra Zeneca, France, 0.5%) and ketamine (25mg) in 0.5 ml (Ketam, EIPICO, Egypt, 50 mg/mL),. Total volume is 2 ml will injected. The control group will receive only intrathecal bupivacaine (7.5 mg) in 1.5 ml plus 0.5ml normal saline to achieve total volume of 2 ml.

Anaesthetic technique

participants will receive oral medication 60 minutes preoperatively with 0.5 mg/kg of midazolam.

After arrival at the OR, an intravenous (IV) 18-20G catheter was placed and infusion of 20 ml/kg NaCl 0.9% will start. Standard monitoring electrocardiogram (ECG), heart rate (HR), oxygen saturation (SpO2), and non-invasive blood pressure (BP) will be started.

Dural puncture was made in the sitting position with a 25 gauge spinal needle using a median approach. After aspiration, the dose of anaesthetic as indicated in the envelope was injected over two minutes. The time of Dural puncture was used as the Primary starting point of assessment. The medications injection will be over 10 s with no barbotage and the needle orifice cephaled. After intrathecal injection, participants will kept sitting for 10 minutes, after that the patient will lie in the lithotomy position and received 100% O2 (4 L/min) with face mask.

Ten minutes after the Dural puncture, participants will asked to lie down and the level of sensory block will tested with an alcohol swab. Motor block was tested by modified Bromage scale (0 = no motor block, 1 = able to flex ankle and bend knees, 2 = able to flex ankle, and 3 = full motor block) [21], and surgery in the supine position will allow to started. In case of failed block, general anaesthesia will be induced.

Non-invasive BP taken every 5 minutes and HR were assessed in the OR. Reduction of mean BP (MAP) and HR >20% from baseline was judged clinically significant. A decrease in systolic BP below 90 mmHg will be treated with 5 mg of IV ephedrine, HR<45 beats per minute (bpm) will be treated with 0.5 mg of IV atropine.

Patient assessment:

* Demographics (age, gender, type of surgery); duration of anesthesia (from the moment of dural puncture until patient left the OR) and surgery in minutes.
* Rate of success (failed block, number of attempts made, ease of performance scale 1-3, where 3 = easy to perform, 2 =moderate, 1 = difficult, multiple attempts needed);
* level of sensory (dermatomes) and motor (Bromage scale) block10 minutes after dural puncture, at the end of surgery, and in the ward every 30 minutes until resolution of the block and afterwards at 6, 9, 12, 18 and 24 hours postoperatively;
* MAP and HR every 5 minutes in the OR, then every 4 hours for postoperative 24 hours;
* Complications during performance of anesthesia: paresthesias, toxic reactions,
* Level of postoperative pain on a written VAS scale (0-10 mm).
* Time of 1st analgesic request, and number of requests for each patient will be recorded in the 1st 24 hours.
* Consumption of rescue analgesia; if VAS is ≥ 5 in the form of 30 mg intramuscular (IM) repeated twice as patient satisfaction and 0.1mg of morphine for up stocking of pain
* Postoperative complications:

  - Urinary retention (0-2 scale, where 0 = normal urination, 1 = difficult spontaneous urination, and 2 = unable to urinate, catheterization needed.
* Postoperative nausea and vomiting (PONV; 0-3 scale, where 0 = no nausea, 1 = slight nausea, 2 = nausea and single vomiting, and 3 = multiple vomiting) [15],
* Postdural puncture headache (PDPH) at day 1 postoperatively and 10 days later by phone call at home,
* Transient neurologic symptoms (TNS), backache, itching, allergic reactions, time of postoperative recovery, time to urinate, duration of sensory and motor block, and time to stand and walk unsupported

Statistical analysis

The data will be recorded on and analyzed using SPSS-12. The results will be presented as Mean ±SD or percent of patients. For proportions, Pearson test or Fisher's test will be used. Student's t-test being used for quantitative variables. A p-value of <0.05 will be considered to show statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included in the study only if they meet all of the following criteria:
* Patients scheduled for perianal surgeries.
* Age 18-55 years.
* ASA physical status I-II.

Exclusion Criteria:

* Subjects will be excluded from the study for any of the following reasons:
* Patient refusal
* Any contraindication of regional anaesthesia
* Failed Technique

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
- Duration of saddle block | 24 hours post-operative
  (time from intrathecal injection to the time of first complain of pain, first request for analgesia, or a reported NRS >4)

SECONDARY OUTCOMES:
Evaluation of the need of supplemental analgesia | 24 hours post-operative
  time of 1st dose

IPD SHARING:
Plan to Share IPD: No